CLINICAL TRIAL: NCT00562198
Title: Effects of Single Doses of Stalevo 200 and Levodopa/Carbidopa 200/50mg on Striatal 11C-Raclopride Binding Potential in Parkinson's Disease Patients With Wearing-Off Symptoms;an Open, Randomised, Active-Controlled,Two-Period Crossover Study.
Brief Title: PET-Study: Effects of Single Doses of Stalevo and Levodopa/Carbidopa on Striatal 11C-Raclopride Binding
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Illogistical results found in interim evaluation.
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Irja Korpela, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2939121
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Parkinson´s Disease
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Investigational drug Stalevo 200
  Interventions: Drug: entacapone and carbidopa; Drug: Sinemet 200mg/50mg

INTERVENTIONS:
Drug: entacapone and carbidopa — Entacapone 200mg carbidopa 50mg
Drug: Sinemet 200mg/50mg — Sinemet 200mg/50mg once

SUMMARY:
This is an open, randomised, active-controlled, 2-period crossover study comparing the effect of single doses of Stalevo 200 and Sinemet on striatal (putamenal and caudate) 11C-raclopride BP in PD patients with wearing-off symptoms. The study consists of 4 visits: a screening visit (visit 1), 2 treatment periods (period 1=visit 2, period 2=visit 3) separated by a minimum wash-out period of at least 3 days, and an end-of-study visit (visit 4). Subjects will be randomly allocated to start the period 1 with a single dose of Stalevo 200 or Sinemet. After the wash-out the study drug on period 2 will be administered according to a crossover design.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with idiopathic Parkinson's disease according to the UK Brain Bank criteria.
2. Predictable wearing-off symptoms with a response to standard release levodopa/carbidopa (200/50 mg)during the levodopa challenge test lasting for a minimum of 1.5 h and a maximum of 4 h.
3. The magnitude of response (peak effect) in the levodopa challenge test is at least 30%. The magnitude of response is defined to be the difference between the baseline score and the lowest UPDRS III score during the levodopa challenge test.
4. Hoehn and Yahr stage of at least 2.0 performed during the "ON" state.
5. Treatment with at least 4 daily doses of levodopa/dopa decarboxylase inhibitor (DDCI) (± entacapone(Comtess® or Stalevo) with total daily levodopa dose in the range of 400-1200mg.
6. Unchanged levodopa/DDCI ± entacapone and other antiparkinsonian medication [dopamine agonists,monoamine oxidase B (MAO-B) inhibitor, amantadine and/or anticholinergics with an approved dose], if any, for at least 2 weeks prior to period I.
7. Written informed consent obtained.
8. Age of 45-80 years, inclusive.

Exclusion Criteria:

1. Secondary or atypical parkinsonism.
2. Patients with any unpredictable "OFF"-periods.
3. Patients with moderate to severe treatment-related peak-dose dyskinesia likely to affect the quality of brain magnetic resonance image (MRI) or positron emission tomography (PET) imaging.
4. Failure to adequately respond to the levodopa (levodopa/carbidopa 200/50 mg) challenge test with the duration of response lasting less than 1.5 h or more than 4 h.
5. Presence of a basal ganglia lesion in the MRI image or any other factor(s) that would make MRI or PET imaging likely to be unsatisfactory.
6. Presence of any ferromagnetic objects that would make brain MRI imaging contraindicated.
7. Patients with a history of laboratory abnormality consistent with, or clinically significant cardiovascular,pulmonary, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness, which may influence the outcome of the study including the interpretation and usage of MRI and PET images for the study purposes.
8. History of neuroleptic malignant syndrome (NMS) and/or non-traumatic rhabdomyolysis, malignant melanoma, narrow-angle glaucoma or pheochromocytoma.
9. Severe hepatic impairment.
10. Any abnormal electrocardiogram (ECG) finding with clinical relevance.
11. Female patients of childbearing potential (menstruating or less than 2 years post-menopausal) if they are not using adequate contraception during the study (defined as hormonal contraception, intrauterine device or surgical sterilization) or female patients who are pregnant or lactating.
12. Treatment with cabergoline.
13. Concomitant treatment with apomorphine, MAO-A inhibitors or non-selective MAO inhibitors.
14. Concomitant treatment with any drugs with antidopaminergic action (e.g. with D2 receptor blocking properties) less than two weeks or within five times the elimination half-life of a given drug prior to the first study drug administration. As an exception, the use of domperidone is allowed.
15. Current, regular use of any iron preparation that cannot be interrupted for the duration of the study
16. Patients who are likely to need a rescue dose of levodopa after the withdrawal from their own levodopa/DDCI ± entacapone medication prior to PET imaging.
17. Known hypersensitivity to active study drug substances or to any of the excipients.
18. Participation in other drug studies within 30 days prior to study entry.
19. Blood donation or loss of significant amount of blood within 60 days prior to the screening.
20. Any other condition that in the opinion of the investigator could create a hazard to the subject safety,endanger the study procedures or interfere with the interpretation of study results.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The difference between the study drugs in change in striatal 11C-raclopride BP.Striatal 11C-raclopride BP will be determined with PET scans performed at baseline and from 2.5 to 3.5 h after the study drug administration. | Post-dosing PET scan

SECONDARY OUTCOMES:
The difference between the study drugs in levodopa mean C2.5- 3.5h. | C 2.5-3.5h

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, Dr, Principal Investigator — Turku PET Centre, Turku, Finland
Locations (5):
- Finland (5):
  - Helsinki University Hospital, Department of Neurology, Helsinki
  - Oulu University Hospital, Department of Neurology, Oulu
  - Porin Lääkäritalo, Pori
  - FinnMedi Tutkimus Oy, Tampere
  - CRST, Turku